CLINICAL TRIAL: NCT06492213
Title: Effectiveness and Safety of Platelet-Rich Plasma Combined With Pulsed Radiofrequency to Treat Patients With Infraorbital Neuralgia
Brief Title: The Efficacy and Safety of Pulsed Radiofrequency Combined With Platelet-rich Plasma for Infraorbital Neuralgia
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Qinghai People's Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Day surgery and Pain Management Affiliation, Beijing Tiantan Hospital
Other Study IDs: KY2023-263-03-03
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Infraorbital Neuralgia; Platelet-rich Plasma
Keywords: Infraorbital neuralgia; platelet- rich plasma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRP+PRF: PRF procedure will be performed at first. Puncture point will be identified at the surface projection point of the infraorbital foramen on the affected side, and after reach the infraorbital foramen under the guidance of thin-slice CT (2 mm/layer, Somaton, Siemens Company, Munich, Germany). The radiofrequency electrode needle (PMK-21-100; Baylis Medical Inc.) will be inserted into the trocar after removal of the the stylet and confirmation of no bleeding or air when withdrawal using a syringe. The standard PRF mode will be initially set at 42℃, then the PRF output voltage will be gradually increased to the highest voltage the patient can tolerate, and the treatment will be continued for 360 seconds. After PRF, the PRF electrode needle will be removed and 2 milliliter PRP will be injected into the same puncture site through the trocar needle.
  Interventions: Other: No interventions
- PRF alone: Puncture point will be identified at the surface projection point of the infraorbital foramen on the affected side, and after reach the infraorbital foramen under the guidance of thin-slice CT (2 mm/layer, Somaton, Siemens Company, Munich, Germany). The radiofrequency electrode needle (PMK-21-100; Baylis Medical Inc.) will be inserted into the trocar after removal of the the stylet and confirmation of no bleeding or air when withdrawal using a syringe. The standard PRF mode will be initially set at 42℃, then the PRF output voltage will be gradually increased to the highest voltage the patient can tolerate, and the treatment will be continued for 360 seconds.
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — It is a observational study to investigate the efficacy and safety of PRP combined PRF on IONa compared to PRF alone.

SUMMARY:
This is a multicenter, prospective, observational, propensity score matching, cohort, and assessor-blinded study designed to compare the effectiveness and safety of PRP injections combined with PRF treatment with PRF alone in patients with IONa who are responded poorly to conventional therapies and are reluctant to receive destructive therapies for seeking a better minimally invasive treatment strategy.

DETAILED DESCRIPTION:
Infraorbital neuralgia (IONa) is one of a rare but devastating type of facial pain and lack of current consensus on the management. Previously, we have proved the efficacy of pulsed radiofrequency (PRF) in treatment of IONa. However, refractory patients have not received more ideal treatment until now. Platelet-rich plasma (PRP), as supraphysiological concentration of platelets, can provide prolonged neuropathic pain relief with almost no complications. To date, the efficacy of PRP combined with PRF in the treatment of IONa has not yet been proved. We will conduct this multicenter, prospective, observational, propensity score matching, cohort, and assessor-blinded study to evaluate the efficacy and safety of PRP combined with PRF in treating refractory IONa patients who were reluctant to receive destructive therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years;
2. Paroxysmal or persistent stabbing pain in the distribution area of the infraorbital nerve and positive response to diagnostic block (1 ml of 2% lidocaine) prior to treatment;
3. NRS score≥7;
4. Scheduled for PRF treatment for IONa；
5. Signed informed consent.

Exclusion Criteria:

1. Platelet count <105*109/L, ongoing anticoagulation therapy or antiplatelets treatment, coagulation disorders or bleeding disorders;
2. Severe cardiopulmonary or hepatorenal dysfunction;
3. Infection at the puncture site; .
4. Neuralgia secondary to tissue damage around the infraorbital foramen from causes such as maxillary sinusitis or tumor;
5. History of destructive treatments such as radiofrequency thermocoagulation, chemical ablation, infraorbital neurectomy, infraorbital nerve avulsion, etc;
6. History of mental disorders；
7. History of narcotic drug abuse;
8. Unable to cooperation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Power Analysis and Sample Size (PASS) V.15.0 software (NCSS Corporation, Kaysville, UT, USA) is used to compute the sample size. The results indicate that a study with a power of 80% and two-sided statistical significance level (alpha) of 0.05 would require 64 participants each group. Considering 10% loss to follow-up and an additional 40% loss after propensity score matching, the total sample size of this study will be 237 patients. And we are planning to enroll 240 patients totally considering the convenience of sample collection and statistics
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The 1-year response rate | 12-month period
  cases responding to treatment/total number of cases*100%

SECONDARY OUTCOMES:
Response rate | at 1 day, 1 week, 1 month, 3 months, 6 months, 9 months, 12 months after operation
  cases responding to treatment/total number of cases*100%
Dosage of carbamazepine | at 1 day, 1 week, 1 month, 3 months, 6 months, 9 months, 12 months after operation
  dosage of carbamazepine
Numeric rating scale (NRS) score of pain | at 1 day, 1 week, 1 month, 3 months, 6 months, 9 months, 12 months after operation
  0 representing no pain and 10 representing the most severe pain imaginable
Patients' quality of life (QOL) | at 1 day, 1 week, 1 month, 3 months, 6 months, 9 months, 12 months after operation
  evaluated by 12-item short-form health survey (SF-12) scores,Response categories vary from 2 to 6 and can be transformed to scale scores ranging from 0 ('the worst') to 100 ('the best')
Patient satisfaction scores (PSS） | at 1 day, 1 week, 1 month, 3 months, 6 months, 9 months, 12 months after operation
  0 point indicates unsatisfactory, while 10 points indicate the most satisfactory
Adverse events (AEs) | at 30minutes, 1 day, 1 week, 1 month, 3 months, 6 months, 9 months, 12 months after treatment.
  such as dizziness, facial swelling, facial ecchymoma, eye injury, infection, etc

CONTACTS AND LOCATIONS:
Overall Officials: Luo Fang, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Fang Luo, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
not yet decided